CLINICAL TRIAL: NCT04317859
Title: Behavioural Activation Therapy for Bipolar Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Zainab Samaan (Zena), Associate Professor, St. Joseph's Healthcare Hamilton
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BRAVE for Bipolar: 5924
Record Dates: First submitted 2020-02-27; First posted 2020-03-23 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Bipolar Disorder
Keywords: Behavioural Activation; Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioural Activation (Intervention) (Experimental): Originally a component of Cognitive Therapy, Behavioural Activation is the use of strategies such as activity scheduling, master/pleasure ratings, and graded task assignments to modify one's perception of specific situations. Behavioural Activation involves the use of activities to improve life situations and mood symptoms.
  Interventions: Behavioral: Behavioural Activation
- Waitlist (Control) (No Intervention): The Control group (waitlist) will receive treatment as usual while waiting to receive BA intervention (at the end of intervention group therapy time, which will consist of 18 sessions over an 14 week period). This group will be assessed by clinical staff that offer treatment as usual for mood symptoms and quality of life measures during the waiting time.

INTERVENTIONS:
Behavioral: Behavioural Activation — Behavioural Activation (BA) is a therapy previously shown to be effective in depressive disorders. This form of therapy involves modification of activities in order to change perceptions of specific situations, thereby improving mood. The BA treatment program will consist of 18 two-hour visits over 14 weeks (twice weekly group visits for the first 8 weeks, followed by two individual visits over 6 weeks).
  Arms: Behavioural Activation (Intervention)

SUMMARY:
Mood disorders including bipolar disorder and depression are common disabling disorders with depression affecting 11.2 to 16.0% of the general population and the lifetime prevalence of bipolar disorders at an estimated 4.4%. Although treatment with antidepressants medications is common and effective in some patients, 42.7% of patients show inadequate response to treatment with antidepressants and a large proportion (55.3%) continue to have ongoing depressive symptoms. Psychological and behavioural interventions such as cognitive behavioural therapy (CBT) and behavioural activation (BA) are effective treatment for depression alone or in combination with antidepressants. Depression can also occur in the context of bipolar disorder which is characterized by recurrent episodes of depression and mania (DSM-5). The depressive episodes within bipolar disorder may be similar to depressive disorder, however the management of these episodes is fraught with the challenge that antidepressant pharmacotherapy may precipitate manic episodes and lead to further destabilization of bipolar disorder. Therefore, an alternative to antidepressants and additional therapies are needed to support patients' recovery and mood stability, as well as to achieve better treatment response and remission. BA is not currently available in a structured format and has not been tested for its effectiveness in bipolar disorders in a specialized hospital-based program. The evidence for BA has been investigated in depression however the evidence for bipolar disorder is lacking, therefore this study aims to assess the effectiveness of BA as treatment for bipolar disorder.

DETAILED DESCRIPTION:
This study is a pragmatic randomized controlled trial to test the effectiveness of behavioural activation in bipolar disorder. The pragmatic randomized controlled trial study design is a parallel 1:1 allocation comparing behavioural activation plus treatment as usual to waitlist control group plus treatment as usual. For this study the investigators will adopt the following principals simulating naturalistic real life clinical setting to test the study question based on the pragmatic design:

No restrictive inclusion criteria will be used. Adults with bipolar disorder will be asked to participate in this study Clinicians will deliver the BA program to participants randomized to receive the intervention The intervention will be an add-on to treatment as usual The comparison group will receive treatment as usual that may include medications, CBT and other therapies as required and decided by their clinical care The primary outcome is clinically relevant (improvement in depressive and manic symptoms)

Both the intervention and control groups will be assessed as intention to treat analysis with no measures to improve adherence to the study intervention or the comparator.

Patients with a diagnosis of bipolar disorders attending the mood disorders clinic, referred for assessment of bipolar disorder at the clinic or referred from community or other hospital services to the mood disorders clinic will be approached for participation in the study. In addition, family practices in the community will be informed of the study and asked to refer directly to the trial. Following initial screening for eligibility, potential participants will be asked to provide written informed consent prior to any study related procedures.

The investigators will employ a parallel group design to evaluate the effects of behavioural activation intervention to improve bipolar disorder-related outcomes. Eligible and consenting patients will be randomly allocated to the intervention or control arms using a 1:1 allocation ratio. Allocations will be generated using the computerized system. The randomization will use a block randomization system of block sizes of 2, 4 and 6. Allocation will be conducted by a research personnel who is not a clinician and will not know the participant clinical status to maintain allocation concealment.

This trial is an open label trial as blinding is not possible for participants (behavioural activation intervention) or the clinician administering the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Bipolar Disorder
* Must be able to provide written informed consent
* Must be able to attend program sessions

Exclusion Criteria:

* Inability to understand written and spoken English
* Primary diagnosis other Bipolar Disorder.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-05-07 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Assess the effectiveness of a structured, therapist administered, group therapy program of Behavioural Activation (BA) in addition to usual care, on depressive symptoms | End of the study period (14 weeks)
  The Beck Depression Inventory (BDI-II) is administered to measure the effectiveness of BA on depressive symptoms. Items in the BDI are scored on a scale of 0-63, where 63 is the maximum score and higher scores are associated with more severe symptoms.
Assess the effectiveness of a structured, therapist administered, group therapy program of Behavioural Activation (BA) in addition to usual care, on manic symptoms | End of the study period (14 weeks)
  The Altman Self-Rating Scale (ASRS) is administered to measure the effectiveness of BA on manic symptoms. The ASRS has 5 items and a maximum score of 20; higher scores are associated with increased severity.

SECONDARY OUTCOMES:
Test the effects of BA on changes in health parameters | End of the study period (14 weeks)
  Quality of Life, as measured by the Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form (Q-LES-Q-SF), Short-Form 12 Health Survey (SF-12), and the Work and Social Adjustment Scale (WSAS). The Q-LES-Q-SF is a 14-item questionnaire scored between 0% and 100%, where higher percentages are indicative of a higher QOL. WSAS scores items between 0 (indicating no impairment) and 8 (indicating severe impairment); total scores greater than 20 indicate severe psychopathology and symptomology. The SF-12 generates two summary scores, the physical component score (PCS) and the mental component score (MCS); scores range between 0 and 100, where 100 is associated with the highest level of health state.
Economic evaluation of the BA program in the study population. | End of the study period (14 weeks)
  Economic evaluation of the BA program will be assessed using the EuroQol 5-Dimension 5-Level (EQ-5D-5L), a commonly used measure of health status and quality of life in a variety of clinical conditions. Each of 5 items are scored between 0 to 4; the maximum score of the EQ-5D-5L is 1, with higher scores being associated with poorer health.

CONTACTS AND LOCATIONS:
Overall Officials: Zainab Samaan, MBChB, PhD, Principal Investigator — St. Joseph's Healthcare Hamilton
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No